CLINICAL TRIAL: NCT07343440
Title: A Randomized Controlled Trial on the Impact of Indirect Calorimetry-Guided Nutritional Support on Patient-Centered Outcomes in Critically Ill Patients - The OPTICal Study
Brief Title: Trial on the Impact of Indirect Calorimetry-Guided Nutritional Support on Patient-Centered Outcomes in Critically Ill Patients - The OPTICal Study
Acronym: OPTICal
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: HEIDEGGER CP (Other)
Collaborators: University Hospital, Zürich (Other); GHOL Nyon Hospital (Unknown)
Responsible Party: Sponsor-Investigator, HEIDEGGER CP, Prof, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: OPTICal2025
Record Dates: First submitted 2025-08-07; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Critical Illness; ICU
Keywords: Nutrition; Indirect calorimetry; Nutrition therapy; Predictive formula
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group - Indirect Calorimetry Group (Experimental)
  Interventions: Other: Indirect Calorimetry Group
- Control Group - Formula-Based Group (Active Comparator)
  Interventions: Other: Control Group - Formula-Based Group

INTERVENTIONS:
Other: Indirect Calorimetry Group — * Nutritional targets measured by IC starting on Day 4
  * Repeated IC measurements 2 times weekly performed with the QNRG+ device
  * Gradual escalation to 80%-100% caloric coverage by Day 4
  Arms: Intervention Group - Indirect Calorimetry Group
Other: Control Group - Formula-Based Group — * Nutritional targets determined using predictive equations (pragmatic, set at local level)
  * Escalation as per local protocol
  Arms: Control Group - Formula-Based Group

SUMMARY:
This multicentric randomized controlled trial aims to evaluate whether indirect calorimetry (IC)-guided nutritional support improves patient-centered outcomes in critically ill adult patients compared to standard formula-based nutritional strategies. The study includes mechanically ventilated patients expected to remain in the ICU for more than 72 hours. The intervention group will receive nutritional targets based on measured resting energy expenditure using the QNRG+ device, with a gradual escalation of energy delivery following current ESPEN guidelines. The primary outcome is quality of life at 3 months post-ICU admission, assessed using the EQ-5D-5L. Secondary outcomes include functional recovery, muscle preservation, infection rates, and rehospitalization. This study is the first to assess the long-term impact of IC-guided nutrition on recovery and quality of life using a patient-centered approach.

ELIGIBILITY:
Inclusion Criteria:

All patients admitted to the ICU with the following criteria:

* ≥18 years old
* On Mechanical Ventilation
* Expected ICU length of stay >72 hours

Exclusion Criteria:

* Refusal of the family or patient
* Patient transferred from another ICU
* Pregnant patient
* Patient is planned for a withdrawal of care or is actively dying
* Cognitive disorder before ICU
* Patient is in jail
* Patients already enrolled in the ongoing NutriPhyT trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 356 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Quality of life (EQ-5D-5L) | At 3 months after ICU admission
  Measured using the EQ-5D-5L: 0-100

SECONDARY OUTCOMES:
Mortality | Up to 3 months after ICU admission
Nosocomial infection | Up to 28 days after ICU admission
  Defined as the initiation of a new antibiotic treatment lasting at least 72 hours, associated with a documented diagnosis of infection in the patient's chart
Pressure soar | Up to 28 days after ICU admission
Energy deficit in kcal | Up to 28 days after ICU admission
  according to the energy target defined by IC or predictive formula depending on the randomization group
Protein deficit in grams | Up to 28 days after ICU admission
  according to the protein target defined by predictive formula
Ventilation-free days | Measured at day 28 after ICU admission
ICU free-days | Measured at day 28 after ICU admission
Functional recovery: Bartel Index | At ICU discharge or up to 28 days after ICU admission and at 3 months after ICU discharge
  Using Barthel Index: 0-100
Gerneral well-being: Edmonton Symptom Assessment Scale | At ICU discharge or up to 28 days after ICU admission and at 3 months after ICU discharge
  Using Edmonton Symptom Assessment Scale (ESAS) : 0-90
Readmission and rehospitalization rates | Until 3-month post-ICU admission
Discharge place | Until 3 months after ICU admission
Return to work | Until 3 months after ICU admission
Disability and functioning: WHO Disability Assessment Schedule | At 3-month post ICU admission
  Using WHO Disability Assessment Schedule (WHODAS 2.0): 0-48
Disability and functioning: Clinical Frailty Scale | At 3-month post ICU admission
  Using Clinical Frailty Scale (CFS): 1-9
Disability and functioning: Short-form 12 | At 3-month post ICU admission
  Using Short-form 12 (SF-12): 0-100
Disability and functioning: MOCA-5 | At 3-month post ICU admission
  Using montreal cognitive assessment- 5 min (MOCA-5): 0-15
Disability and functioning: Patient Health Questionnaire-9 | At 3-month post ICU admission
  Using Patient Health Questionnaire-9 (PHQ-9): 0-27

CONTACTS AND LOCATIONS:
Locations (3):
- Switzerland (3):
  - Geneva University Hospital, Geneva
  - GHOL, Nyon
  - Zürich University Hospitals, Zurich

IPD SHARING:
Plan to Share IPD: Undecided